CLINICAL TRIAL: NCT06651827
Title: Clinical Evaluation of the Effectiveness of the Er:Cr:YSGG Laser in Reducing Dentin Sensitivity: A Cross-Sectional Study
Brief Title: Clinical Evaluation of the Effectiveness of the Er:Cr:YSGG Laser in Reducing Dentin Sensitivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Can Tho University of Medicine and Pharmacy (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Vo Xuan Quang
Record Dates: First submitted 2024-10-19; First posted 2024-10-22 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2023-06

CONDITIONS: Dentin Sensitivity
Keywords: Dentin hypersensitivity; Er,Cr:YSSG laser; Yeaple Probe; Visual Analog Scale
MeSH Terms: conditions — Dentin Sensitivity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dentin sensitivity was measured before and after treatment (Experimental): Dentin sensitivity was measured using the Yeaple Probe and air stimulation tests before and after treatment
  Interventions: Diagnostic Test: Dentin sensitivity was measured using the Yeaple Probe and air stimulation tests before and after treatment

INTERVENTIONS:
Diagnostic Test: Dentin sensitivity was measured using the Yeaple Probe and air stimulation tests before and after treatment — Dentin sensitivity was measured using the Yeaple Probe and air stimulation tests before and after treatment. The effectiveness of the treatment was assessed at baseline, 30 minutes, 1 week, and 1 month post-treatment using the Visual Analog Scale (VAS) and Yeaple Probe scores.

SUMMARY:
This study aims to evaluate the clinical effectiveness of the Er:Cr laser in reducing dentin hypersensitivity (DH), a common dental condition characterized by sharp pain in response to thermal, mechanical, chemical, or osmotic stimuli.

DETAILED DESCRIPTION:
Dentin Hypersensitivity is one of the common and uncomfortable clinical issues for patients, characterized by sharp pain when the dentinal tubules are stimulated by thermal, mechanical, chemical, or osmotic agents. This sensitivity often appears in the canine and premolar areas, particularly in the cervical third of the tooth surface. The main cause of DH is dentin exposure, which occurs when the enamel or cementum covering the root surface is lost, usually due to factors such as improper brushing techniques, erosion-induced abrasion, or harmful habits like bruxism. Dentin exposure can also occur due to periodontal disease, gingival recession, or periodontal interventions, such as root planing. One of the most widely accepted theories explaining the mechanism of DH is the hydrodynamic theory proposed by Brännström in 1984. According to this theory, when the dentinal tubules are exposed, pressure changes in the surrounding tissue cause fluid movement within the tubules, stimulating mechanoreceptors in the pulpal nerves, resulting in sharp pain. The diagnosis and treatment of DH are complex due to its multifactorial nature, requiring thorough examination to rule out other oral pathologies and ensure the health of the pulp and gingiva.

Various treatment methods for DH have been proposed in the literature, ranging from modifying brushing habits, guiding patients on diet, occlusal adjustment, to using desensitizing agents such as potassium nitrate, potassium oxalate, and calcium phosphate. Some approaches also involve using bonding systems, adhesive materials, or even lasers to occlude the dentinal tubules and reduce sensitivity. In recent years, the use of dental lasers as an alternative treatment for DH has gained significant attention from researchers. Commonly used lasers include high-power lasers such as Nd:YAG, Er:YAG, Er,Cr:YSGG… as well as low-power lasers in photobiomodulation therapy. The Er,Cr:YSGG laser is of particular interest due to their operation at a wavelength of 2780 nm, which is highly absorbed by water. This allows for the evaporation of fluid in the dentinal tubules, leaving insoluble salts that help seal the tubules and reduce sensitivity symptoms. According to a study by Yilmaz et al. (2011), the Er,Cr:YSGG laser not only provides rapid relief but also maintains its effect for up to three months without causing significant side effects.

Due to the subjective nature of DH, assessing the level of sensitivity is often challenging. However, measurement tools such as the Visual Analog Scale VAS or Yeaple pressure probe have been used in studies to provide more reliable measurement results. The objective of this study is to evaluate the effectiveness of the Er,Cr:YSGG laser in the treatment of DH.

ELIGIBILITY:
Inclusion Criteria:

* Patients >18 years old
* Express a desire for treatment for their dentin hypersensitivity
* Only sensitive teeth without indications for restorative procedures were considered eligible
* Informed consent was obtained from all participants

Exclusion Criteria:

- Patients with underlying systemic conditions or those taking medications that could affect the study outcomes, such as analgesics, anti-inflammatory drugs, or sedatives within 72 hours prior to enrollment

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2023-06-15 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-15 (Actual)

PRIMARY OUTCOMES:
The objective of this study is to evaluate the effectiveness of the Er,Cr:YSGG laser in the treatment of Dentin Sensitivity | Dentin sensitivity was measured using the Yeaple Probe and air stimulation tests before of the Er,Cr:YSGG laser in the and after treatment.
  The objective of this study is to evaluate the effectiveness of Dentin Sensitivity using the Yeaple Probe

CONTACTS AND LOCATIONS:
Overall Officials: Quang Xuan Vo, Principal Investigator — Can Tho University of Medicine and Pharmacy
Locations (1):
- Can Tho University of Medicine and Pharmacy, Can Tho, Vietnam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Haneet RK, Vandana LK. Prevalence of dentinal hypersensitivity and study of associated factors: a cross-sectional study based on the general dental population of Davangere, Karnataka, India. Int Dent J. 2016 Feb;66(1):49-57. doi: 10.1111/idj.12206. Epub 2015 Nov 19. PMID 26582076
- [Result] Yilmaz N, Baltaci E, Baygin O, Tuzuner T, Ozkaya S, Canakci A. Effect of the usage of Er,Cr:YSGG laser with and without different remineralization agents on the enamel erosion of primary teeth. Lasers Med Sci. 2020 Sep;35(7):1607-1620. doi: 10.1007/s10103-020-03015-0. Epub 2020 May 29. PMID 32472426